CLINICAL TRIAL: NCT05633498
Title: The Effect of a Self-help Book for Shift Work Related Problems - a Randomized Controlled Trial
Brief Title: Self-help Book for Shift Work Related Problems
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bergen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HEWOS_RCT_SWD2022
Record Dates: First submitted 2022-11-21; First posted 2022-12-01 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Shift-work Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-help book (Experimental): A self-help book for coping with shift work
  Interventions: Other: Book
- Sleep hygiene advice (Active Comparator): A sheet of paper with basic and standard sleep hygiene advice
  Interventions: Other: Sleep hygiene

INTERVENTIONS:
Other: Book — Self-help book describing advice to cope with shift work
  Arms: Self-help book
Other: Sleep hygiene — Basic sleep hygiene advice on a piece of paper
  Arms: Sleep hygiene advice

SUMMARY:
The aim is to assess whether a self-help book for coping with shift work will reduce complaints in relation to shift work.

DETAILED DESCRIPTION:
This study is a randomized controlled trial evaluating the effect of a self-help book for shift work related problems compared to the effect of sleep hygiene advice in participants with shift work disorder. 300 participants will be randomized to receive either the book or the sleep hygiene advice. Participants complete questionnaires about sleep, sleepiness and health at baseline and after 6 months after receiving the written material. The main aims are to assess whether the book is more effective to reduce sleep and sleepiness problems in relation to shift work, and to reduce the prevalence of shift work disorder, to increase knowledge about sleep and circadian rhythms, improve health, and reduce turnover intention.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms suggesting shift work disorder
* Health care worker

Exclusion Criteria:

* Below 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-11-18 (Actual); Primary Completion 2025-03-18 (Estimated); Study Completion 2025-03-18 (Estimated)

PRIMARY OUTCOMES:
Sleep problems | 6 months
  Self-reported sleep problems in relation to shift work on a validated scale - Bergen Shift Work Sleep Questionnaire (BSWSQ). Questions range from 0 to 4 with higher values indicating more sleep problems.
Sleepiness problems | 6 months
  Self-reported sleepiness in relation to shift work on a validated scale - Bergen Shift Work Sleep Questionnaire (BSWSQ). Questions range from 0 to 4 with higher values indicating more sleepiness.

SECONDARY OUTCOMES:
Shift work disorder | 6 months
  Prevalence of shift work disorder based on international criteria
Knowledge about shift work and health | 6 months
  Questions about sleep, circadian rhythms and shift work
Sick leave | 6 months
  Self-reported sickness absence
Turnover intention | 6 months
  Self-reported turnover intention on a validated scale (TI) with scores ranging from 0 to 4 with higher values indicating more turnover intention.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Bergen, Bergen, Hordaland, Norway

IPD SHARING:
Plan to Share IPD: No